CLINICAL TRIAL: NCT03451136
Title: Value of Third Trimester Cervical Length Measurement in Predicting Risk and Severity if Antepartum Haemorrhage in Cases of Placenta Previa
Brief Title: Cervical Length in Cases of Placenta Previa
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Mahmoud Eid, Ass.prof obs&Gyn., Cairo University
Other Study IDs: Cairo university obgyn 14534
Record Dates: First submitted 2018-02-05; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Placenta Previa
Keywords: Placenta previa; Cervical length; Antepartum haemorrhage
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study establishes the relationship between cervical length and whether it can be used to predict haemorrhage and preterm delivery in cases of placenta previa.

DETAILED DESCRIPTION:
Some studies have reported an association between ultrasonographic decreased cervical length and the likelihood of complications as antepartum or post-partum haemorrhage requiring an emergency caesarean section (CS) .

The safety of trans-vaginal scanning is not in doubt, and the technique now has widespread acceptance. As a consequence, the clinical presentation of placenta previa has changed and most low lying placentas are diagnosed during the second trimester anomaly scan.

The objective of this study was to establish if there is a relation between transvaginal ultrasonographic measurement of cervical length in cases of placenta previa and whether it can be used as a predictor for antepartum haemorrhage or not.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-45 years old
2. Single Pregnancy
3. Fetal gestational age 28 to < 36 weeks
4. Normal amniotic fluid index (AFI)
5. Diagnosis of placenta previa by pelvic ultrasound that was confirmed when the lower placental edge overlies the internal cervical os on transvaginal ultrasound (TVS).

Exclusion Criteria:

1. Threatened preterm labor and maternal use of vaginal progesterone.
2. Preterm premature rupture of membranes;
3. Polyhydramnios;
4. Presence of cercelage and history of cervical cone biopsy which both affect cervical length.
5. Diagnosis of multiple fetal anomalies;
6. Women with other risk factors for intra-partum hemorrhage

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant females aged between 25-40 years
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-15 (Estimated)

PRIMARY OUTCOMES:
Cervical length measured in mm in relation to antepartum haemorrhage | 4 months
  To find out the relationship between cervical length measured by transvaginal ultrasound and occurrence of antepartum hemorrhage in cases of placenta previa.

SECONDARY OUTCOMES:
Need for blood transfusion | 4 months
  Yes or no and no.of packed units
Need for caesarean hysterectomy | 4 months
  Yes or no
Type of cesarean delivery | 4 months
  Elective or emergency cesarean delivery
Need for neonatal ICU | 4 months
  Yes or no